CLINICAL TRIAL: NCT00723190
Title: An Open-Label, Chronic Exposure Evaluation of the Safety of CLONICEL (Clonidine HCl Sustained Release) in the Treatment of Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Open-Label, Chronic Exposure, Safety Study of CLONICEL (Clonidine HCl Sustained Release) in Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Shionogi Clinical Trials Administrator, Shionogi
Organization: Shionogi Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLON-303
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Results first posted 2012-02-27 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: CLONICEL; Attention Deficit Hyperactivity Disorder; clonidine HCl sustained release
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): CLONICEL (Clonidine HCl sustained release)
  Interventions: Drug: CLONICEL (Clonidine HCl sustained release)

INTERVENTIONS:
Drug: CLONICEL (Clonidine HCl sustained release) — 0.1 mg for 1 week; the dose may be escalated to 0.2 mg/day at week 2, 0.3 mg/day at week 3, and 0.4 mg/day at week 4

SUMMARY:
The purpose of this 12-month, multi-center, open-label study is to evaluate the safety of CLONICEL (clonidine HCl sustained release) when administered chronically under regular clinical conditions either as monotherapy or in combination with stimulant therapy to children and adolescents with attention deficit hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject who has completed either study CLON-301 or study CLON-302, or discontinued early for reasons other than adverse events necessitating discontinuation
* Age between 6 and 17 years, inclusive
* Diagnosis of attention deficit hyperactivity disorder of the hyperactive or combined inattentive/hyperactive subtypes according to Diagnostic and Statistical Manual of Mental Disorders IV (DSM IV) criteria
* General good health as judged by the Principal Investigator
* Body mass index (BMI) ≥ 5th percentile of the subject's age group according to the CDC growth chart. BMI is calculated using the formula: weight (kg) / [height (m)]2
* Subject as well as parent/guardian able to sign informed assent or consent form

Exclusion Criteria:

* If female of child-bearing potential, pregnant or lactating or does not agree to use a medically acceptable form of birth control, such as hormonal medication, double-barrier method, or intrauterine device
* Presence of a clinically significant illness or abnormality on physical examination or clinical laboratory evaluations that, in the opinion of the investigator, would increase the safety risks from clonidine administration or interfere with the ability of the patient to take part in the study.
* Presence of clinically significant abnormality on centrally interpreted electrocardiogram readings
* History or presence of a concomitant psychiatric disorder requiring psychotropic medication or a severe concomitant axis I or axis II disorder that could interfere with study assessments in the judgment of the Principal Investigator
* Presence of a disorder that would interfere with the absorption, metabolism, or excretion of clonidine
* Presence of alcohol or drug abuse.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2008-01; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (26):
- United States (26):
  - Little Rock, Arkansas
  - El Centro, California
  - Irvine, California
  - San Diego, California
  - Bradenton, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Lauderhill, Florida
  - Miami, Florida
  - Orlando, Florida
  - Bardstown, Kentucky
  - Baltimore, Maryland
  - Rochester Hills, Michigan
  - St Louis, Missouri
  - Voorhees Township, New Jersey
  - Willingboro, New Jersey
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Houston, Texas
  - Lake Jackson, Texas
  - Wharton, Texas
  - Clinton, Utah
  - Kirkland, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 27 study centers in the United States. First subject visit was on January 09, 2008 and last subject completed the study on March 08, 2010
Pre-assignment Details: Candidates enrolled in this study (CLON-303) were subjects who completed studies using KAPVAY (CLONICEL) as add-on therapy with stimulants (CLON-302) and as monotherapy (CLON-301). There was no screening period for this study. The safety follow-up visit from these two prior studies (CLON-301 and CLON-302) was the baseline visit for current study
Groups:
- KAPVAY (CLONICEL): One tablet (0.1 mg) for 1 week; At Week 2, one additional 0.1 mg tablet; At Week 3, one additional 0.1 mg tablet; At Week 4, one last 0.1 mg tablet bringing the total dose to a maximum of 0.4 mg/day (0.2 mg twice daily)
Period: Overall Study
Arm/Group | KAPVAY (CLONICEL)
Started | 303 (Study CLON-301 (168 participants) and Study CLON-302 (135 participants))
SAFETY POPULATION | 301
Completed | 161 (53 participants completed 6-month protocol and 108 participants completed 12-month protocol)
Not Completed | 142
Not completed — Withdrawal by Subject | 45
Not completed — Lost to Follow-up | 37
Not completed — Adverse Event | 18
Not completed — Lack of Efficacy | 16
Not completed — Protocol Violation | 15
Not completed — Other-Premature Discontinuation | 9
Not completed — Other-Not included in safety population | 2

BASELINE CHARACTERISTICS:
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.1 (2.75)
Age, Continuous [Median (Full Range); unit: Years] | 10.0 [6.0 to 17.0]
Age, Customized [Number; unit: Participants]
  6-12 Years | 239
  > 12-17 Years | 62
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristics are presented for the subjects in the safety population (total 301 participants)
  Participants
    Female | 80
    Male | 221
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 186
  Black/African American | 69
  Hispanic or Latino | 25
  Other | 21
Weight [Mean (Standard Deviation); unit: Kilograms] — Data collected from 291 participants
  Kilograms | 42.3 (18.94)
Weight [Median (Full Range); unit: Kilograms] — Data collected from 291 participants
  Kilograms | 38.1 [19.6 to 131.0]

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessment in Terms of Adverse Events (Treatment-emergent [TEAEs] and Serious [SAEs])
Description: Safety assessments were performed at each study visit according to the time and events schedule. All safety analyses were based on safety population
Time Frame: 1 year
Population: The analysis of the safety data was performed for the safety population which included subjects who took one or more doses of study medication. All subjects in the trial are included in the safety population
Measure: Number; unit: Participants
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 301
Participants
  Total Safety Population | 301
  Subjects with ≥1 TEAEs | 246
  Subjects with ≥1 related TEAEs | 178
  Subjects with ≥1 SAEs | 2
  Subjects with ≥1 TEAEs leading to discontinuation | 17

2. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHDRS-IV Scale) (18 Items Scored, 0 [Never/Rarely] to 3 [Very Often]; Total Possible Score Range, 0-54) at Months 1, 2, 3, 4, 6, 9, and 12
Description: The ADHDRS-IV consists of 18 items designed to reflect symptoms of ADHD. Each item is scored on a scale of 0 (Never or rarely) to 3 (Very Often). The subscales of the ADHDRS-IV included the Inattention and the hyperactivity/Impulsivity subscales (total possible score range, 0-54). The Inattention subscale consists of the sum of 9 items: 1, 3, 5, 7, 9, 11, 13, 15, and 17. The Hyperactivity/Impulsivity subscale consists of the sum of 9 items: 2, 4, 6, 8, 10, 12, 14, 16, and 18
Time Frame: At baseline, months 1, 2, 3, 4, 6, 9, and 12
Population: Efficacy summaries and analyses are based on the efficacy evaluable population which included subjects who took one or more doses of study medication and had at least one post-baseline efficacy measurement
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 290
Units on a scale
  1-month (n = 229) | -13.7 (11.52)
  2-month (n = 221) | -14.4 (11.73)
  3-month (n = 203) | -14.8 (12.55)
  4-month (n = 142) | -16.3 (12.59)
  6-month (n = 184) | -14.6 (12.04)
  9-month (n = 119) | -18.1 (12.66)
  12-month (n = 98) | -14.6 (14.05)

3. Primary Outcome: Safety Assessment in Terms of Adverse Events (Treatment-emergent [TEAEs] and Serious [SAEs])
Description: Safety assessments were performed at each study visit according to the time and events schedule. All safety analysis were based on safety population
Time Frame: 1 year
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 301
Events
  Total number of TEAEs | 954
  Total number of related TEAEs | 438
  Total number of SAEs | 2

4. Primary Outcome: Change From Baseline in 12-lead Electrocardiogram in Terms of QT, QTc Fridericia (QTcF), and QTc Bazett's (QTcB) at Week 4
Time Frame: At baseline and at Week 4
Population: Data was analyzed based on safety population which included subjects who took one or more doses of study medication. All subjects in the trial are included in the safety population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 280
milliseconds
  QT | 17.9 (25.69)
  QTcF | 1.4 (16.42)
  QTcB | -8.0 (22.15)

5. Primary Outcome: Change From Baseline in Body Weight at Weeks 1, 2, 3, 4, and Months 2, 3, 4, 5, 6, 9, and 12
Time Frame: At baseline and at weeks 1, 2, 3, 4, and months 2, 3, 4, 5, 6, 9, and 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 301
Kilograms
  week 1 (n = 283) | 0.3 (2.25)
  week 2 (n = 283) | 0.4 (2.28)
  week 3 (n = 278) | 0.6 (2.39)
  week 4 (n = 269) | 0.7 (2.42)
  month 2 (n = 246) | 0.9 (2.61)
  month 3 (n = 232) | 1.2 (2.97)
  month 4 (n = 212) | 1.4 (3.25)
  month 5 (n = 47) | 1.7 (5.63)
  month 6 (n = 204) | 2.1 (3.84)
  month 9 (n = 123) | 3.6 (3.72)
  month 12 (n = 123) | 4.5 (4.83)

6. Primary Outcome: Change From Baseline in Diastolic Blood Pressure at Week 4
Description: Blood pressure was measured with the subject in a sitting position and resting for at least 2 minutes prior to taking the measurement. The dominant arm was used for the measurement
Time Frame: At baseline and at Week 4
Population: Data was anlyzed based on safety population which included subjects who took one or more doses of study medication. All subjects in the trial are included in the safety population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 277
mmHg | -4.2 (9.13)

7. Primary Outcome: Change From Baseline in Systolic Blood Pressure at Week 4
Description: as for outcome 6
Time Frame: At baseline and at Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 277
mmHg | -5.0 (10.71)

8. Primary Outcome: Change From Baseline in Body Temperature at Week 4
Description: Temperature was measured with the subject in a sitting position and resting for at least 2 minutes prior to taking the measurement
Time Frame: At baseline and at Week 4
Population: Data analysis was performed on safety population which included subjects who took one or more doses of study medication. All subjects in the trial are included in the safety population
Measure: Mean (Standard Deviation); unit: Fahrenheit
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 278
Fahrenheit | -0.08 (0.791)

9. Primary Outcome: Change From Baseline in Heart Rate at Week 4
Description: Heart rate was measured with the subject in a sitting position and resting for at least 2 minutes prior to taking the measurement
Time Frame: At baseline and at Week 4
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 277
beats per minute | -7.0 (13.59)

10. Primary Outcome: Change From Baseline in 12-lead Electrocardiogram in Terms of Heart Rate at Week 4
Time Frame: At baseline and at Week 4
Population: Data analysis involved the safety population which included subjects who took one or more doses of study medication. All subjects in the trial are included in the safety population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 280
beats per minute | -10.6 (14.32)

11. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) at Months 1, 2, 3, 4, 6, 9, and 12
Description: CGI-S scale:
  1 = Normal, not ill at all; 2 = Borderline ill; 3 = Mildly ill; 4 = Moderately ill; 5 = Markedly ill; 6 = Severely ill; 7 = Among the most extremely ill patients
Time Frame: At baseline, months 1, 2, 3, 4, 6, 9, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 301
Units on a scale
  1-month (n = 229) | -1.2 (1.17)
  2-month (n = 220) | -1.3 (1.12)
  3-month (n = 202) | -1.3 (1.29)
  4-month (n = 143) | -1.5 (1.19)
  6-month (n = 185) | -1.4 (1.15)
  9-month (n = 119) | -1.7 (1.35)
  12-month (n = 97) | -1.4 (1.46)

12. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Improvement (CGI-I) at Months 1, 2, 3, 4, 6, 9, and 12
Description: CGI-I scale:
  1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse
Time Frame: At baseline, months 1, 2, 3, 4, 6, 9, and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | KAPVAY (CLONICEL)
Number analyzed (Participants) | 301
Units on a scale
  1-month (n = 229) | 2.5 (1.05)
  2-month (n = 220) | 2.5 (1.11)
  3-month (n = 202) | 2.5 (1.10)
  4-month (n = 143) | 2.3 (1.04)
  6-month (n = 185) | 2.4 (1.11)
  9-month (n = 119) | 2.1 (1.11)
  12-month (n = 97) | 2.4 (1.39)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | KAPVAY (CLONICEL)
Serious Adverse Events (participants affected / at risk) | 2/301
Other Adverse Events (participants affected / at risk) | 246/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KAPVAY (CLONICEL) (N=301)
Suicidal Behavior (Psychiatric disorders) | 1
Cellulitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KAPVAY (CLONICEL) (N=301)
Somnolence (Psychiatric disorders) | 96
Affect Lability (Psychiatric disorders) | 12
Emotional Disorder (Psychiatric disorders) | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 37
Vomiting (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 12
Diarrhoea (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 8
Upper Respiratory Tract Infection (Infections and infestations) | 39
Gastroenteritis Viral (Infections and infestations) | 20
Nasopharyngitis (Infections and infestations) | 10
Headache (Nervous system disorders) | 49
Insomnia (Nervous system disorders) | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 18
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 16
Influenza (Respiratory, thoracic and mediastinal disorders) | 8
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 6
Fatigue (General disorders) | 37
Irritability (General disorders) | 28
Body Temperature Increased (Investigations) | 22
Weight Increased (Investigations) | 11
Decreased Appetite (Metabolism and nutrition disorders) | 25
Rhinitis Seasonal (Immune system disorders) | 7
Dermatitis Contact (Immune system disorders) | 6
Dizziness (Cardiac disorders) | 9
Hand Fracture (Injury, poisoning and procedural complications) | 6
Otitis Media Acute (Ear and labyrinth disorders) | 6
Rash (Skin and subcutaneous tissue disorders) | 6

LIMITATIONS AND CAVEATS:
Efficacy results need to be reviewed in the context that the study is an open-label/non-placebo controlled study. No formal statistical testing of efficacy results has been done. No adjustments have been made to account for drop-outs or missing data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.